CLINICAL TRIAL: NCT01455467
Title: A Prospective Evaluation of Open-angle Glaucoma Subjects on One Topical Hypotensive Medication Randomized to Treatment With One or Two Trabecular Micro-bypass Stents in Conjunction With Cataract Surgery
Brief Title: Open-angle Glaucoma Subjects on One Topical Hypotensive Medication Randomized to Treatment With One or Two Trabecular Micro-bypass Stents in Conjunction With Cataract Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Glaukos Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GCF-024
Record Dates: First submitted 2011-09-28; First posted 2011-10-20 (Estimated); Last update posted 2022-08-31 (Actual); Status verified 2022-08

CONDITIONS: Open-angle Glaucoma
Keywords: Open angle glaucoma; Pigmentary glaucoma; Pseudoexfoliative glaucoma
MeSH Terms: conditions — Glaucoma, Open-Angle

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- One iStent (Active Comparator): Implantation of one iStent in conjunction with cataract surgery
  Interventions: Device: One iStent
- Two iStent (Active Comparator): Implantation of two iStent devices in conjunction with cataract surgery
  Interventions: Device: Two iStent

INTERVENTIONS:
Device: One iStent — Implantation of one iStent in conjunction with cataract surgery
  Arms: One iStent
Device: Two iStent — Implantation of two iStent in conjunction with cataract surgery
  Arms: Two iStent

SUMMARY:
Evaluation of intraocular pressure (IOP) lowering effect of one iStent versus two iStents in conjunction with cataract surgery in subjects with primary open-angle glaucoma, washed out of one anti-glaucoma medication prior to stent implantation.

ELIGIBILITY:
Inclusion Criteria:

* Phakic study eye requiring cataract removal and posterior chamber intraocular lens (PC-IOL) implantation
* Primary open-angle glaucoma (including pigmentary or pseudoexfoliative)

Exclusion Criteria:

* Aphakic or pseudophakic with posterior or anterior chamber IOLs (PC-IOLs or AC-IOLs) (study eye)
* Prior stent implantations (study eye)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2011-09 (Actual); Primary Completion 2019-10-18 (Actual); Study Completion 2019-10-18 (Actual)

PRIMARY OUTCOMES:
Mean diurnal IOP reduction of ≥ 20% vs. baseline mean diurnal IOP | 12 Months

CONTACTS AND LOCATIONS:
Overall Officials: Lilit A Voskanyan, MD, PhD, Principal Investigator — S.V. Malayan Ophthalmological Center, Yerevan, Armenia
Locations (1):
- S.V. Malayan Ophthalmological Center, Yerevan, Armenia